CLINICAL TRIAL: NCT01077466
Title: Natalizumab Treatment of Progressive Multiple Sclerosis
Acronym: NAPMS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Copenhagen University Hospital, Hvidovre (Other); Biogen (Industry); University of Copenhagen (Other); Signifikans ApS (Other)
Responsible Party: Principal Investigator, Finn Sellebjerg, Assoc. professor, MD, PhD, DMSci, Finn Sellebjerg, Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NAPMS version 3.4
Record Dates: First submitted 2010-02-26; First posted 2010-03-01 (Estimated); Last update posted 2012-02-17 (Estimated); Status verified 2012-02

CONDITIONS: Primary Progressive Multiple Sclerosis; Secondary Progressive Multiple Sclerosis
Keywords: Primary Progressive Multiple Sclerosis; Secondary Progressive Multiple Sclerosis; Natalizumab; Treatment; Safety; Efficacy; Cerebrospinal fluid; Osteopontin
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive | interventions — Natalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Natalizumab (Experimental): 24 patients: 12 with secondary progressive multiple sclerosis 12 with primary progressive multiple sclerosis
  Interventions: Drug: Natalizumab

INTERVENTIONS:
Drug: Natalizumab — 300 mg Natalizumab IV for every 4 week for 56 weeks (15 doses for every patient)
  Other Names: Tysabri

SUMMARY:
The purpose of this study is to study safety and efficacy of natalizumab treatment of primary and secondary progressive multiple sclerosis.

This will be done by measuring the effect of treatment on inflammation in the CNS by means of osteopontin levels in the cerebrospinal fluid (CSF). Safety measures further includes physical and neurological examination,blood samples and MRI measures of disease activity.

DETAILED DESCRIPTION:
The study will include 12 secondary progressive multiple sclerosis patients and 12 primary progressive multiple sclerosis patients to treatment with IV natalizumab for 60 weeks. At baseline and week 60 a lumbar puncture will be performed. MRI scans will be performed at baseline week 12 and week 60.Safety blood samples will be collected every 12 week.

ELIGIBILITY:
Inclusion Criteria:

* Age between 19 and 55 years
* Progressive disease course of multiple sclerosis (primary or secondary)
* Duration of progressive phase of at least 1 year
* Progression of > 1 EDSS point during the last 2 years (>½ EDSS point if EDSS > 5,5)
* EDSS </= 6.5
* Written and informed consent

Exclusion Criteria:

* Pregnancy, breast-feeding or lack of anti.conception for fertile women.
* Attack during the last month before inclusion.
* Treatment with methylprednisolone during 3 months before inclusion.
* Treatment with interferon-beta, glatirameracetate, immunoglobulin G or other immune-modulating treatment 3 months prior to inclusion.
* Treatment with mitoxantrone, cyclophosphamide, azathioprine or other strong immunosuppressive drug 6 months prior to inclusion.
* Prior experimental treatment with strong immunosuppressive drug which the treating physician means will influence the results of the trial.
* Diseases associated with immunodeficiency.
* Treatment with other anticoagulant than aspirin.
* Current malign disease.
* Diabetes Mellitus or other autoimmune disease.
* Renal insufficiency or creatinine > 150 μmol/l.
* Travel in tropical areas 3 months prior to inclusion.
* Acute or chronic infectious diseases, which the treating physician finds relevant (e.g.hepatitis B virus, hepatitis C virus, HIV).
* Psychiatric disease or other circumstances that may limit the patients participation in the trial.
* Contraindication for MRI scan or gadolinium contrast .
* Known hypersensitivity to natalizumab.

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2010-03; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Cerebrospinal fluid (CSF) osteopontin | Change from baseline to week 60
  The primary endpoint is change in CSF osteopontin from baseline to week 60.

SECONDARY OUTCOMES:
Expanded disability status scale (EDSS) | Baseline to week 60
  Change in expanded disability status scale (EDSS)from baseline to week 60
Timed 25-foot Walk (T25FW) | Baseline to week 60
Multiple Sclerosis Impairment Score (MSIS) | Baseline to week 60
Multiple Sclerosis Functional Composite | Baseline to week 60
Short Form 36 Health Survey (SF36) | Baseline to week 60
CSF Neurofilament Heavy Chain | Baseline to week 60
  Change in neurofilament heavy chain in the cerebrospinal fluid
CSF Myelin Basic Protein | Baseline to week 60
  Change in myelin basic protein in CSF from baseline to week 60
Atrophy | Week 12 to week 60
  Change in normalised brain volume (NBV), grey matter volume (GMV) og white matter volume (WMV) from week 12 to week 60
Magnetization transfer ratio (MTR) | Baseline to week 60
  Change in MTR in whole brain, lesions, normal-appearing grey matter (NAGM) og normal-appearing white matter (NAWM) from baseline to week 60
Diffusion transfer imaging (DTI) | Baseline to week 60
  Change in FA and ADC in lesions, GM and NAWM between baseline and week 60.
CSF cell count | Baseline to week 60
  Change in CSF cell count from baseline to week 60
Change in IgG-index | Baseline to week 60
CSF nitrogen oxide metabolites | Baseline to week 60
CSF-serum albumine concentration quotient | Baseline to week 60
CSF CXCL13 | Baseline to week 60
Matrix metalloproteinase-9 (MMP-9) | Baseline to week 60
New Gadolinium-enhancing lesions (GdEL) | Baseline to week 60
Volume of lesions on T2-weighted MRI images | Baseline to week 60
Number of new or enlarging lesions on T2-weighted MRI images | Baseline to week 60

CONTACTS AND LOCATIONS:
Overall Officials: Finn Sellebjerg, MD PhD DMSc, Principal Investigator — Danish Multiple Sclerosis Center
Locations (1):
- Danish Multiple Sclerosis Center, Section 2082, Rigshospitalet, Copenhagen, Denmark